CLINICAL TRIAL: NCT05738200
Title: Use of Nordic Hamstring Exercise to Improve Hamstrings Function in Patients After ACL Reconstruction
Brief Title: Nordic Hamstring Exercise After ACL Reconstruction Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toledo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202737
Record Dates: First submitted 2022-11-02; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: ACL Injury; Muscle Weakness; Neuromuscular Manifestations
Keywords: Eccentric exercise; Hamstrings
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Muscle Weakness; Neuromuscular Manifestations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nordic Hamstring Exercise (Experimental): A 4-week (10 session), progressive, Nordic Hamstring Exercise (NHE) protocol will be used for this study.
  Interventions: Other: Nordic Hamstring Exercise
- Control (No Intervention): Patients randomized to the control group will be instructed to avoid any changes to their normal routine (e.g., physical activity level, strength training, etc.). An investigator not involved in data collection will communicate with patients in the control group on a weekly basis to ensure they have not changed their physical activity level and do not have any questions. Patients randomized to the control group will participate in a minimum of 2 study visits at baseline and 4 weeks. These individuals will have the option to open enroll in the intervention group at the completion of their original 4-week study period. Those who choose to enroll in the intervention group at this time will return for 11 additional visits to complete the NHE protocol (visits 3-12) and final assessment (visit 13)

INTERVENTIONS:
Other: Nordic Hamstring Exercise — A 4-week (10 session), progressive, NHE protocol will be used for this study. Immediately following the completion of study visit 1, patients will be informed about the nature of the NHE protocol. Those available and willing to participate will be randomized to an intervention group (NHE, control). Patients randomized to NHE will receive formal instruction about how to correctly perform the exercise, and will be asked to perform several repetitions to familiarize themselves with the exercise and verify proper technique. At this time, patients will be dismissed from study visit 1, and return visits 2-11 will be scheduled to complete the NHE protocol. Patients will return for a final study visit (12) to record post-intervention measurements within 7 days of completing the NHE protocol. A minimum of 48 hours will be used to separate study visits. To accurately assess patients' ability to perform the NHE, all exercise will be performed on a NordBord Hamstring Testing System.
  Arms: Nordic Hamstring Exercise

SUMMARY:
Anterior cruciate ligament (ACL) injuries constitute a significant portion of major knee joint injuries sustained by young, active individuals, and significantly increase risk for long-term disability. Yet the recommended solution to restore joint stability following injury--ACL reconstruction (ACLR)--does not prevent post-traumatic knee osteoarthritis (PTOA). Post-traumatic quadriceps (dys)function is a hallmark characteristic following ACLR, reported to accelerate the onset of PTOA after ACL injury, making the recovery of muscle function a primary concern to clinicians. However, hamstrings muscle function is drastically underrepresented relative to the quadriceps in the context of recovery from ACLR, which impedes the ability to develop targeted treatment approaches. Persistent hamstrings weakness is widely reported in patients who undergo ACLR with a hamstring tendon (HT) autograft, which increases ACL strain, and may contribute to higher graft failure rates in this population. To effectively treat muscular impairments, underlying neuromuscular adaptations known to occur in response to ACLR must be targeted. Eccentric exercise is uniquely suited to enhance neuromuscular function. The Nordic hamstring exercise (NHE) is a specific form of eccentric exercise that is clinically relevant and easy to implement, but has not been explored as an intervention for hamstrings neuromuscular dysfunction in patients who undergo ACLR with HT. To establish an evidence-based treatment model, the investigators will use a single-blind, randomized controlled clinical trial to establish the feasibility and efficacy of a 4-week NHE protocol in patients who undergo ACLR with HT. Separate factorial ANOVAs will be used to assess the effects of group (NHE, control) and time (baseline, 4 weeks) on selected outcomes. Effect sizes will be calculated for within- and between-group comparisons. The investigators expect to observe improvements in hamstrings neuromuscular function following the NHE protocol, and that those improvements will be greater than the control group. Additionally, the investigators expect the protocol to be feasible in terms of intervention adherence and patient retention. This study will identify specific barriers to the implementation of NHE in patients who undergo ACLR with HT, and will provide support for the application of an easy to implement clinical intervention able to address a complex neurophysiological problem.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-35
* History of primary, unilateral ACL reconstruction (ACLR) with hamstrings tendon autograft

Exclusion Criteria:

* Lower extremity orthopedic surgery prior to ACLR
* Post-surgical complication (e.g. infection, delayed healing)
* Multiple ligament knee injury
* Treated articular cartilage lesion
* Known history of knee osteoarthritis
* Concussion within 6 months
* History of neurological disorder
* Currently taking prescription medication that may alter neural excitability (e.g. stimulants, depressants)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2018-07-07 (Actual); Primary Completion 2022-07-13 (Actual); Study Completion 2022-07-13 (Actual)

PRIMARY OUTCOMES:
Change in peak eccentric torque | Baseline, 4 weeks
  Hamstrings
Change in peak isometric torque | Baseline, 4 weeks
  Hamstrings
Change in peak isokinetic torque | Baseline, 4 weeks
  Hamstrings

SECONDARY OUTCOMES:
Change in rate of torque development | Baseline, 4 weeks
  Hamstrings
Change in torque coefficient of variation | Baseline, 4 weeks
  Hamstrings
Change in central activation ratio | Baseline, 4 weeks
  Hamstrings
Change in single leg hop | Baseline, 4 weeks
  Hop for distance
Change in active motor threshold | Baseline, 4 weeks
  Transcranial magnetic stimulation (TMS) derived outcome in semitendinosus
Change in cortical silent period | Baseline, 4 weeks
  Transcranial magnetic stimulation (TMS) derived outcome in semitendinosus
Change in short-interval cortical inhibition | Baseline, 4 weeks
  Transcranial magnetic stimulation (TMS) derived outcome in semitendinosus
Change in intracortical facilitation | Baseline, 4 weeks
  Transcranial magnetic stimulation (TMS) derived outcome in semitendinosus

OTHER OUTCOMES:
Change in visual analog scale | Baseline, 4 weeks
  Current knee pain questionnaire (range: 0 [no pain] to 10 [high pain])
Change in Tampa Scale of Kinesiophobia 11-item | Baseline, 4 weeks
  Fear of pain-related movement and reinjury questionnaire (range: 11 [low fear] to 44 [high fear])
Change in ACL Return to Sport after Injury | Baseline, 4 weeks
  Psychological readiness questionnaire (range: 0 [low readiness] to 100 [high readiness])
Change in International Knee Documentation Committee Subjective Knee Evaluation | Baseline, 4 weeks
  Subjective knee function questionnaire (range: 0 [low function] to 100 [high function])
Change in Knee Injury and Osteoarthritis Outcome Score | Baseline, 4 weeks
  Subjective knee function questionnaire (range: 0 [low function] to 100 [high function])
Veterans RAND 12-Item Health Survey | Baseline, 4 weeks
  Global health questionnaire (range: 0 [low global health] to 100 [high global health])
Change in Tegner Activity Scale | Baseline, 4 weeks
  Subjective activity level questionnaire (range: 0 [low activity] to 10 [high activity])
Change in International Physical Activity Questionnaire | Baseline, 4 weeks
  Subjective activity level (higher values = higher activity level)
Time spent in moderate-to-vigorous physical activity | 4 weeks
  Objectively monitored physical activity
Global Rating of Change | 4 weeks
  Subjective perception of change in knee function following intervention (range: -7 [worse knee function] to 7 [better knee function])
Intrinsic Motivation Inventory | 4 weeks (intervention group only)
  Interest/enjoyment and value/usefulness subscale questionnaires (range: 7 [no interest/enjoyment or value/usefulness] to 49 [high interest/enjoyment or value/usefulness])
Average rating of perceived exertion | 4 weeks (intervention group only)
  Subjective perception of effort/difficulty during exercise questionnaire (range: 6 [light effort] to 20 [high effort]), completed during each intervention session
Average visual analog scale | 4 weeks (intervention group only)
  Average pain or discomfort questionnaire (range: 0 [no pain/discomfort] to 10 [high pain/discomfort]), completed during each intervention session

CONTACTS AND LOCATIONS:
Overall Officials: Grant Norte, PhD, ATC, Principal Investigator — The University of Toledo
Locations (1):
- The University of Toledo, Toledo, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Norte GE, Glaviano NR, Sherman DA, Rush JL, Murray AM. Four-week Nordic hamstring exercise intervention for individuals with ACL reconstruction via hamstrings tendon autograft: feasibility of a pilot randomized controlled trial. Pilot Feasibility Stud. 2025 Apr 3;11(1):37. doi: 10.1186/s40814-025-01624-6. PMID 40181441